CLINICAL TRIAL: NCT00367042
Title: Prospective Study To Determine Whether Tissue Scoring Results In Noticeable Marks Following Mohs Micrographic Surgery
Brief Title: Study to Determine if Tissue Scored With a Scalpel Results in Any Noticeable Marks
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 200513516-1
Record Dates: First submitted 2006-08-19; First posted 2006-08-22 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (No Intervention)
  Interventions: Device: Scalpel for tissue scoring; Device: Surgical marker for tissue marking

INTERVENTIONS:
Device: Scalpel for tissue scoring — During Mohs surgery we will compare the outcomes of scarring, to determine whether a mark (with a pen) or a score with a scalpel will receive the best scar.
Device: Surgical marker for tissue marking — You will be asked to participate, examined, discuss participation have procedure and come in for follow up for photos and check up.

SUMMARY:
Mohs Micrographic Surgery is a well established method for treatment of cutaneous malignancies. Part of this technique requires marking skin surrounding the tumor. There are two ways of marking the tissue, lightly scoring it with a scalpel or marking it with a surgical marker.

This study is to determine if there is a noticeable difference in outcome between patients who have their tissue lightly scored with a scalpel or marked with a surgical marking pen.

DETAILED DESCRIPTION:
Mohs Micrographic Surgery is a well established method utilizing microscopic margin controlled excision for treatment of cutaneous malignancies (See Appendix A). It has the highest cure rate of any of the methods used to treat common cutaneous malignancies and is a proven safe outpatient procedure. Part of the technique requires marking skin surrounding the tumor to correspond with tissue that has been removed and divided into pieces for processing and microscopic examination. Currently there are two established ways of marking the tissue; lightly scoring it with a scalpel or marking it with a surgical marker. Scoring tissue is faster, more accurate, and there is no risk of having the marking washed or rubbed away.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are able to legally consent to study and are scheduled for Mohs Micrographic Surgery to remove their malignancies

Exclusion Criteria:

* Patients who are unable to legally consent themselves, do not wish to participate or who are not scheduled to undergo Mohs Micrographic Surgery.
* Children, those with mental handicaps, pregnant women, prisoners, those with cognitive impairments, and life-threatening diseases will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2005-07; Primary Completion 2006-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The goal of the study is to determine if there are any noticeable differences in outcomes between patients who have their skin scored and those who have their skin marked with a surgical marking pen | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eisen, MD, Principal Investigator — University of California, Davis; Thomas King, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Medical Center Department of Dermatology, Sacramento, California, United States

REFERENCES:
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical